CLINICAL TRIAL: NCT07098052
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Efficacy, and Pharmacokinetics of HDM2020 (FGFR2b-ADC) in Patients With Advanced Solid Tumors
Brief Title: A Study of HDM2020 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HDM2020-101
Record Dates: First submitted 2025-07-18; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HDM 2020 (Experimental): HDM2020
  Interventions: Drug: HDM2020

INTERVENTIONS:
Drug: HDM2020 — FGFR2b-ADC

SUMMARY:
The goal of this clinical trial is to learn if the study drug can work in advanced cancer patients. The main questions it aims to answer are:

* Is the drug safe and tolerable ?
* Does the drug exhibit antitumor activity ?

Participants will receive the study drug once every three weeks, and imaging-based efficacy assessments will be performed every six weeks.

DETAILED DESCRIPTION:
Target population are patients with FGFR2-expressing solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who understand and voluntarily (or legal guardian) sign a written ICF approved by the Institutional Review Board or Independent Ethics Committee.
2. Male or female participants aged ≥18 years.
3. Participants must be patients with advanced or metastatic malignant solid tumors confirmed by histology or cytology, and have experienced sufficient standard treatment failure, or are intolerant to standard treatment, or have no effective standard treatment.
4. Tumor tissue samples are required to be sent to the central laboratory for IHC testing.
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) is 0 or 1.
6. The expected survival time is >3 months.
7. According to the RECIST v1.1, participants in Phase Ia must have at least one evaluable lesion, and participants in Phases Ib must have at least one measurable lesion.
8. Laboratory test results during the screening period indicate that the participants have good organ function.
9. Women of childbearing potential (WOCBP) must be willing to use two appropriate barrier methods of contraception from the time of signing informed consent until 7 months after the last dose of study treatment or use barrier contraception plus hormonal contraception to prevent pregnancy, or abstain from heterosexual intercourse throughout the study period; male participants must agree to take adequate contraceptive measures from the first dose of study treatment until 7 months after the last dose of study treatment.
10. Participants with the willingness and ability to complete regular visits, treatment plans, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Participants with prior treatment with an ADC containing a topoisomerase I (Top I) inhibitor.
2. Participants with active or chronic corneal disorders, history of corneal transplant, keratitis, keratoconjunctivitis, keratopathy, corneal abrasion, inflammation or ulcer, other active eye disorders, and any clinically significant corneal disorders.
3. Participants underwent major surgery within 4 weeks before the first dose; Participants received bone marrow or extensive radiotherapy within 4 weeks before the first dose; received local radiotherapy within 2 weeks before the first dose of the study drug; Participants continuously received systemic corticosteroids; Participants received standard chemotherapy, biological therapy, immunotherapies, any investigational medicinal product (IMP) and other systemic anti-tumor treatments within 4 weeks before the first dose.
4. Participants with active malignant tumors within the past 2 years.
5. Participants not recovered (recovered to ≤ Grade 1 or baseline) from relevant AEs resulting from prior treatments or other anti-cancer therapies.
6. Participants with known active central nervous system (CNS) metastases.
7. Participants with any of the following cardiovascular/cerebrovascular diseases/symptoms/indications: a) Mean resting QTc : ≥470 ms, ECG QTc measured three times within 10 min as the mean value; or those have a history or family history of congenital long QT syndrome; b) Any clinically significant abnormalities in resting ECG in rhythm, conduction, or morphology; c) Left ventricular ejection fraction (LVEF) <50%; d) Participants with a history of myocardial contraction decreased and exhibited related symptoms within 6 months before study drug administration; e) Hypertension uncontrolled by drug therapy
8. At screening, participants with active syphilis, immunodeficiency disease (HIV), active hepatitis B virus (HBV), or active hepatitis C virus (HCV).
9. Presence of interstitial pneumonia, history of idiopathic pulmonary fibrosis, history of organising pneumonia, history of drug-induced pneumonia, history of idiopathic pneumonia, or evidence of active pneumonia found on chest computed tomography (CT) scan during the screening period; prior use of steroid pulse therapy due to pneumonia; Moderate or severe chronic obstructive pulmonary disease (COPD); Pulmonary malignant lymphangitis.
10. Other diseases that may affect the efficacy and safety of the study drug, including but not limited to: a) Active infection requiring antibiotic therapy occurring within 2 weeks prior to the administration of study drug; b) Active autoimmune diseases or a history of autoimmune diseases; c) History of primary immunodeficiency; d) Active pulmonary tuberculosis; e) Participants who have had a clinically significant haemorrhage or significant haemorrhagic diathesis within 4 weeks before signing the informed consent; f) Any severe or uncontrolled systemic disease.
11. Large amounts or symptomatic moderate amounts of pleural effusion, pericardial effusion, or ascites during the screening period, and still poorly controlled after treatments.
12. Unstable thrombosis events requiring therapeutic intervention within 6 months before screening.
13. A history of solid organ transplant.
14. Known or suspected hypersensitivity to the study drug or its analogues.
15. Pregnant and breastfeeding women.
16. The investigator considers that the participant is not suitable to participate in this study.
17. Participants who have received strong CYP3A4 inhibitors within 1 week before dosing, or are expected to require long-term use of strong CYP3A4 inhibitors during the study intervention period and within 30 days after the last dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-11 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerance dose (MTD) of HDM2020 | DLT will be evaluated on 21 days of observation period
  Maximum-tolerated dose (MTD) was defined as the dose level at which the estimated toxicity probability is closest to the target toxicity probability during the dose-escalation phase, within the DLT observation period (21 days) following the first administration of the IMP.
Incidence of Treatment-Emergent Adverse Events | Estimated 1 year
  Incidence rates of adverse events (AE), serious adverse events (SAE)

SECONDARY OUTCOMES:
Time to peak (Tmax) | Estimated 1 year
  Tmax of HDM2020, total antibody, and exatecan will be measured
Half-life time (t1/2) | Estimated 1 year
  t1/2 of HDM2020, total antibody, and exatecan will be measured
Peak Plasma Concentration (Cmax) | Estimated 1 year
  Cmax of HDM2020, total antibody, and exatecan will be measured
Area under the plasma concentration versus time curve (AUC) | Estimated 1 year
  AUC of HDM2020, total antibody, and exatecan will be measured
Objective response rate (ORR) | Estimated 1 year
  Objective response rate (ORR) assessed based on RECIST v1.1 criterion
Duration of response (DoR) | Estimated 1 year
  Duration of response (DoR) assessed based on RECIST v1.1 criterion
Disease control rate (DCR) | Estimated 1 year
  Disease control rate (DCR) assessed based on RECIST v1.1 criterion
Progression-free survival (PFS) | Estimated 1 year
  Progression-free survival (PFS) assessed based on RECIST v1.1 criterion
Overall survival (OS) | Estimated 1 year
  Overall survival (OS) of 6-months and 12-months

OTHER OUTCOMES:
Target expression levels | Estimated 1 year
  Target expression levels and their correlation with antitumor activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No